CLINICAL TRIAL: NCT06847295
Title: Epidural Electrical Stimulation for Motor and Functional Recovery in Patients With Chronic Paralysis Due to Spinal Cord Injury: A Prospective Study Evaluating Gait Restoration, Spasticity Reduction, Pain Management, and Quality of Life Improvements Through Neuromodulation and Intensive Rehabilitation
Brief Title: Epidural Electrical Stimulation to Restore Standing and Walking in Patients With Chronic Paralysis Due to Spinal Cord Injury: A Study on Motor Recovery, Spasticity Reduction, and Quality of Life Improvement Through Neuromodulation and Intensive Rehabilitation
Acronym: EPISTIM-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30702520.6.0000.0068
Record Dates: First submitted 2025-02-18; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries (SCI); Paralysis, Lower Limbs
Keywords: Spinal Cord Injury; Spinal Cord Stimulation; Epidural Stimulation; Neuroplasticity; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Epidural Electrical Stimulation + Intensive Rehabilitation Arm (Experimental): Patients enrolled in this arm will undergo surgical implantation of an epidural spinal cord stimulator (Medtronic Specify 5-6-5 paddle lead and Intellis pulse generator) followed by a 12-month intensive rehabilitation program. After a one-month post-operative recovery period, electrical stimulation will be activated during five supervised physiotherapy sessions per week. The intervention combines neuromodulation with targeted motor and balance exercises to facilitate gait recovery, reduce spasticity, alleviate pain, and enhance overall quality of life. Outcomes will be monitored through clinical scales, surface electromyography, and video documentation, with patients serving as their own controls by comparing pre- and post-implantation performance.
  Interventions: Procedure: Epidural Electrical Stimulation (EES) using an implanted paddle lead and pulse generator combined with a 12-month intensive rehabilitation program.

INTERVENTIONS:
Procedure: Epidural Electrical Stimulation (EES) using an implanted paddle lead and pulse generator combined with a 12-month intensive rehabilitation program. — The intervention consists of surgical implantation of an epidural electrical stimulator using a paddle lead (Medtronic Specify 5-6-5) placed in the lumbar epidural space and a subcutaneously implanted pulse generator (Medtronic Intellis). After a one-month recovery and device calibration period, the stimulator is activated during a 12-month intensive rehabilitation program. Patients receive electrical stimulation during five supervised physiotherapy sessions per week. Stimulation parameters-including pulse width, frequency, and amplitude-are individually optimized based on intraoperative neurophysiological monitoring and ongoing clinical assessments, with the goal of enhancing gait recovery, reducing spasticity, and improving overall motor function and quality of life.

SUMMARY:
Spinal cord injury (SCI) is a major cause of morbidity and disability worldwide, significantly impacting patients' quality of life and functional independence. Despite advances in rehabilitation therapies, many individuals with SCI remain unable to stand or walk. Epidural electrical stimulation (EES) has emerged as a promising neuromodulation therapy to restore motor function in individuals with chronic paralysis.

This prospective clinical study aims to evaluate the efficacy and safety of EES in patients with chronic SCI who have lost the ability to stand or walk. The primary objective is to assess late-stage gait recovery following the implantation of an epidural spinal cord stimulator, using validated clinical scales such as the Fugl-Meyer Assessment - Lower Extremity (FMA-LE) and BMCA VRI.

Secondary objectives include evaluating:

The ability to stand independently (measured by the Berg Balance Scale). Improvements in walking capacity, with or without assistance. Changes in spasticity induced by EES (Modified Ashworth Scale). Reduction in pain perception (DN4, Brief Pain Inventory [BPI], Pain Disability Index [PDI]).

Improvements in neurogenic bladder and bowel dysfunction (NBSS and NBDS). Enhancements in quality of life (SCI-QOL, WHOQOL-BREF) and mood (Beck Depression Inventory [BDI]).

The study will recruit 10 adult patients (ages 18-50) with chronic, stable SCI (≥6 months post-injury) classified as ASIA A or B, with lesions between C7 and T10 and intact segmental reflexes below the injury level. Participants will undergo an intensive 3-month pre-implant rehabilitation program to maximize their baseline motor potential.

Following this period, eligible patients will receive surgical implantation of an epidural spinal cord stimulator (Medtronic Specify 5-6-5 paddle lead and Intellis pulse generator). After a 1-month post-surgical recovery period, patients will engage in a 12-month intensive rehabilitation protocol (5 supervised sessions per week), with the stimulator activated to facilitate motor recovery.

Patients will be assessed monthly through clinical evaluations and surface electromyography (EMG) to measure motor control improvements. Outcomes will be compared before and after EES implantation to determine the effectiveness of the intervention.

This study seeks to provide further evidence on the potential of epidural electrical stimulation in restoring standing and walking abilities in individuals with SCI. If successful, it could contribute to expanding treatment options for patients with chronic paralysis.

DETAILED DESCRIPTION:
Introduction and Rationale:

Spinal cord injury (SCI) is a major cause of long-term disability and diminished quality of life, with current rehabilitation methods often falling short of restoring independent mobility. Emerging evidence suggests that neuromodulation, particularly Epidural Electrical Stimulation (EES), can facilitate the reactivation of dormant spinal networks, thereby promoting motor recovery. Preclinical studies and initial clinical reports have demonstrated that EES can enhance neuroplasticity and improve gait function in patients with chronic paralysis. This study is designed to build on these findings by evaluating the efficacy and safety of EES in a cohort of patients with chronic, stable SCI who have lost the ability to stand or walk.

Study Objectives:

The primary objective of this prospective study is to assess late-stage gait recovery after the surgical implantation of an epidural spinal cord stimulator. Secondary objectives include improvements in standing balance, walking capacity (with or without assistance), reduction in spasticity, pain management, and enhancements in neurogenic bladder and bowel function, as well as overall quality of life and mood. This extended description outlines the technical aspects of the study design, surgical procedure, rehabilitation protocols, and neurophysiological assessments.

Study Design and Overall Methodology:

This is a single-arm, prospective clinical study designed to follow each patient as their own control by comparing pre-operative and post-operative functional status. The study will enroll 10 adult patients with chronic SCI (≥6 months post-injury) classified as ASIA A or B, with lesions located between C7 and T10 and preserved segmental reflexes below the level of injury. Prior to surgical intervention, participants will undergo a 3-month intensive rehabilitation program aimed at maximizing their baseline motor function. This phase includes five supervised physiotherapy sessions per week, during which comprehensive clinical assessments, video documentation, and surface electromyography (EMG) recordings are collected.

Surgical Procedure and Device Implantation:

Following the pre-operative rehabilitation phase, patients will undergo a surgical procedure for the implantation of an epidural spinal cord stimulator. The procedure is performed in a sterile operating room at the Hospital das Clínicas, Faculty of Medicine, University of São Paulo. Key technical details of the procedure include:

Patient Positioning and Preparation: Patients are positioned prone, and the operative site is marked using fluoroscopic guidance. Standard aseptic protocols are followed.

Incision and Exposure: A midline skin incision, approximately 5-8 cm in length, is made between the T12 and L2 vertebral levels. Dissection is carried out through the subcutaneous tissue and paravertebral muscles.

Creation of an Interlaminar Window: An interlaminar window is created at the L1/L2 level to provide access to the epidural space.

Electrode Implantation: A paddle lead (Medtronic Specify 5-6-5, featuring 16 channels arranged in three rows) is implanted in the lumbar epidural space, targeting the region between T11 and L1 to cover the dermatomes from L1 to S2. Intraoperative neurophysiological monitoring using EMG is employed to verify the precise placement of the electrode.

Pulse Generator Placement: A subcutaneous pocket is created in the right flank for the implantation of the pulse generator (Medtronic Intellis). The device is tested intraoperatively to ensure optimal performance and appropriate neuromodulatory response.

Post-Operative and Rehabilitation Protocol:

After a post-surgical recovery period of one month-allowing for wound healing and initial device programming-patients will enter the post-implant rehabilitation phase. This phase consists of a 12-month period during which patients participate in intensive, supervised physiotherapy sessions (five sessions per week). During these sessions:

Activation of EES: The epidural electrical stimulation is activated to facilitate motor recovery. Stimulation parameters (e.g., intensity, frequency, pulse width) are individually adjusted based on patient response and neurophysiological feedback.

Ongoing Evaluations: Regular assessments are conducted monthly using both clinical scales and surface EMG recordings. These evaluations monitor improvements in gait, balance, and overall motor control. Video recordings are also made to document functional performance.

Neurophysiological and Technical Assessments:

A critical component of the study is the use of surface electromyography (EMG) to provide quantitative measures of muscle activity and neuromuscular coordination. Technical details include:

Equipment: A wireless 8-channel EMG system (Trigno Avanti Research+, Delsys) will be used for data acquisition.

Muscle Groups Monitored: EMG electrodes will be placed on key muscles involved in gait and posture, including the iliopsoas, vastus lateralis, rectus femoris, tibialis anterior, semitendinosus, gastrocnemius, soleus, extensor hallucis longus, biceps femoris, and gluteus maximus.

Data Acquisition: EMG signals are filtered (band-pass range between 30 and 500 Hz) and digitized at a sampling rate of 2 kHz. Data analysis is performed offline using Matlab (R2019a) to correlate neuromuscular responses with clinical outcomes.

Safety and Risk Management:

The safety profile of EES is well established in the literature. However, potential risks include surgical complications such as infection, hematoma, device migration, or transient worsening of neurological status. To mitigate these risks, the study incorporates:

Intraoperative Monitoring: Continuous EMG monitoring during electrode implantation to ensure proper placement.

Post-Operative Care: Close monitoring during the recovery phase and strict adherence to infection control protocols.

Adverse Event Reporting: All complications will be recorded and managed according to established clinical guidelines.

Study Timeline and Follow-Up:

The overall study duration for each participant is approximately 16 months, which includes:

A 3-month pre-operative rehabilitation phase. Surgical implantation of the EES device. A 1-month post-operative recovery period. A 12-month post-implant rehabilitation and evaluation phase. Regular follow-up visits will be scheduled for clinical assessments, EMG recordings, and video documentation to continuously monitor progress and adjust therapy as needed.

Ethical Considerations and Regulatory Compliance:

The study protocol has been approved by the Ethics Committee for Research Project Analysis at Hospital das Clínicas, Faculty of Medicine, University of São Paulo (HC-FMUSP). All participants will provide written informed consent prior to enrollment. Given the significant unmet need for effective treatments in chronic SCI and the promising results of neuromodulation in preliminary studies, the design of this study-with patients serving as their own control-is considered ethically justifiable. The study complies with institutional, national, and international regulatory guidelines regarding clinical research and device implantation.

Significance and Expected Impact:

This study aims to provide robust evidence on the efficacy of epidural electrical stimulation in promoting functional motor recovery in patients with chronic spinal cord injury. By combining advanced neuromodulatory techniques with intensive rehabilitation, the study seeks to demonstrate improvements in gait, balance, and overall quality of life. Successful outcomes could lead to broader clinical application of EES and represent a significant advancement in the management of chronic SCI.

Conclusion:

The proposed study is a comprehensive investigation into the application of epidural electrical stimulation as a therapeutic intervention for chronic spinal cord injury. Through meticulous surgical technique, rigorous rehabilitation protocols, and detailed neurophysiological assessments, the study is designed to explore the mechanisms of neuromodulation and validate the clinical benefits of EES. The integration of technical and clinical data is expected to contribute valuable insights that may ultimately transform the treatment landscape for patients with severe, chronic paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 50 years.
* Stable spinal cord injury (SCI) at least 6 months post-injury.
* Classified as ASIA A or B with inability to stand or walk.
* Injury located between C7 and T10.
* Intact segmental reflexes below the level of injury.
* Ability to understand and sign the informed consent form.
* Willingness and capability to attend daily physiotherapy sessions.
* Clinically stable overall health as determined by the investigators.

Exclusion Criteria:

* Current use of electronic devices such as baclofen pumps or cardiac pacemakers.
* Presence of comorbidities that increase surgical risk (e.g., anticoagulation therapy, cardiopulmonary issues).
* Locomotor deformities or additional neurological disorders that may compromise evaluation.
* Significant dysautonomia or history of stroke or myocardial infarction associated with autonomic dysreflexia.
* MRI evidence of complete spinal cord transection, significant spinal atrophy, or significant syringomyelia.
* Uncontrolled pain, severe spasticity, or other conditions that hinder rehabilitation participation.
* Suspected abuse of opioids, alcohol, or other illegal substances.
* Estimated life expectancy of less than 2 years due to severe concomitant malignant or clinical conditions.
* Clinically significant mental health disorders.
* Botulinum toxin injections received in the past 6 months.
* Presence of voluntary movements during EMG testing in the lower extremities.
* Unhealed vertebral fractures.
* Presence of pressure ulcers.
* Active infection.
* Pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Late-Stage Gait Recovery Assessed by the Fugl-Meyer Assessment for Lower Extremities | Baseline and monthly evaluations over 12 months following epidural stimulator implantation
  Evaluates lower limb motor function using the Fugl-Meyer Assessment for Lower Extremities (0-86 points; higher scores indicate better function). Baseline measurements taken before epidural stimulator implantation
Late-Stage Gait Recovery Assessed by the Brain Motor Control Assessment - Voluntary Response Index | Baseline and monthly evaluations over 12 months following epidural stimulator implantation
  Evaluates voluntary motor control and coordination using the Brain Motor Control Assessment - Voluntary Response Index (0-100 points; higher scores indicate improved control). Baseline measurements taken pre-implantation

SECONDARY OUTCOMES:
Balance Assessed by the Berg Balance Scale | Baseline and monthly evaluations over 12 months post-implantation
  Measures balance performance using the Berg Balance Scale (0-56 points; higher scores indicate better balance). Baseline assessments conducted prior to intervention
Walking Ability | Baseline and monthly evaluations over 12 months post-implantation
  Assesses the ability to walk with or without assistance as a dichotomous outcome (able versus not able). Baseline status recorded before intervention
Spasticity Assessed by the Modified Ashworth Scale | Baseline and monthly evaluations over 12 months post-implantation
  Quantifies muscle tone using the Modified Ashworth Scale (0-4 scale; higher scores indicate greater spasticity). Baseline evaluations performed pre-implantation
Pain Perception Assessed by the Douleur Neuropathique 4 Questions | Baseline and monthly evaluations over 12 months post-implantation
  Evaluates neuropathic pain intensity using the Douleur Neuropathique 4 Questions (0-10 scale; higher scores indicate greater pain). Baseline assessments conducted pre-intervention
Pain Severity Assessed by the Brief Pain Inventory | Baseline and monthly evaluations over 12 months post-implantation
  Measures pain severity using the Brief Pain Inventory. Baseline assessments recorded before intervention
Pain-Related Disability Assessed by the Pain Disability Index | Baseline and monthly evaluations over 12 months post-implantation
  Quantifies disability due to pain using the Pain Disability Index (0-70 scale; higher scores indicate greater disability). Baseline evaluations performed pre-implantation
Neurogenic Bladder Function Assessed by the Neurogenic Bladder Symptom Score | Baseline and monthly evaluations over 12 months post-implantation
  Evaluates bladder dysfunction using the Neurogenic Bladder Symptom Score. Baseline measurements taken pre-intervention
Neurogenic Bowel Function Assessed by the Neurogenic Bowel Dysfunction Score | Baseline and monthly evaluations over 12 months post-implantation
  Assesses bowel dysfunction using the Neurogenic Bowel Dysfunction Score (0-47 scale; higher scores indicate more severe dysfunction). Baseline evaluations recorded before intervention
Quality of Life Assessed by the World Health Organization Quality of Life - Brief Version | Baseline and monthly evaluations over 12 months post-implantation
  Measures quality of life using the World Health Organization Quality of Life - Brief Version. Baseline assessments conducted before intervention
Mood Assessed by the Beck Depression Inventory | Baseline and monthly evaluations over 12 months post-implantation
  Evaluates depressive symptoms using the Beck Depression Inventory (0-63 scale; higher scores indicate more severe depression). Baseline assessments conducted pre-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Alves Lepski, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified individual participant data (IPD) that underlies all published results. Shared IPD will include baseline demographic data, detailed clinical outcomes (e.g., FMA-LE and BMCA VRI scores), secondary outcome measures (balance, ambulation, spasticity, pain levels, bladder/bowel function, quality of life, and mood assessments), and neurophysiological data such as surface electromyography recordings and video documentation. This comprehensive dataset will be made available upon reasonable request via a secure, password-protected repository, enabling replication and further research. All data will be anonymized in compliance with applicable privacy regulations to ensure participant confidentiality and data integrity.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The individual participant data (IPD) will be made available starting 6 months after the publication of the primary study results. The data will remain accessible for a period of 5 years from the start of availability. Researchers can request access to the de-identified IPD via a secure, password-protected repository, with all requests reviewed for compliance with privacy regulations and data sharing agreements.
Access Criteria: The de-identified individual participant data (IPD) will be shared with qualified researchers, healthcare professionals, and institutions for legitimate scientific, educational, or health-related purposes. To request access, individuals must submit a formal application outlining their research objectives and intended analyses, including plans for data security and confidentiality. Requests will be reviewed by the study steering committee, which will assess the scientific merit of the proposed research, its alignment with the study's goals, and compliance with ethical standards. IPD will be shared through a secure, password-protected repository, with access granted only to those who meet all criteria.

REFERENCES:
- [Background] Angeli CA, Edgerton VR, Gerasimenko YP, Harkema SJ. Altering spinal cord excitability enables voluntary movements after chronic complete paralysis in humans. Brain. 2014 May;137(Pt 5):1394-409. doi: 10.1093/brain/awu038. Epub 2014 Apr 8. PMID 24713270
- [Background] Krogh K, Christensen P, Sabroe S, Laurberg S. Neurogenic bowel dysfunction score. Spinal Cord. 2006 Oct;44(10):625-31. doi: 10.1038/sj.sc.3101887. Epub 2005 Dec 13. PMID 16344850
- [Background] The World Health Organization Quality of Life assessment (WHOQOL): position paper from the World Health Organization. Soc Sci Med. 1995 Nov;41(10):1403-9. doi: 10.1016/0277-9536(95)00112-k. PMID 8560308
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Pollard CA. Preliminary validity study of the pain disability index. Percept Mot Skills. 1984 Dec;59(3):974. doi: 10.2466/pms.1984.59.3.974. No abstract available. PMID 6240632
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Hallett M. NINDS myotatic reflex scale. Neurology. 1993 Dec;43(12):2723. doi: 10.1212/wnl.43.12.2723. No abstract available. PMID 7802740
- [Background] Angeli C, Rejc E, Boakye M, Herrity A, Mesbah S, Hubscher C, Forrest G, Harkema S. Targeted Selection of Stimulation Parameters for Restoration of Motor and Autonomic Function in Individuals With Spinal Cord Injury. Neuromodulation. 2024 Jun;27(4):645-660. doi: 10.1016/j.neurom.2023.03.014. Epub 2023 May 4. PMID 37140522
- [Background] Ditunno PL, Patrick M, Stineman M, Ditunno JF. Who wants to walk? Preferences for recovery after SCI: a longitudinal and cross-sectional study. Spinal Cord. 2008 Jul;46(7):500-6. doi: 10.1038/sj.sc.3102172. Epub 2008 Jan 22. PMID 18209742
- [Background] GBD 2016 Traumatic Brain Injury and Spinal Cord Injury Collaborators. Global, regional, and national burden of traumatic brain injury and spinal cord injury, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 Jan;18(1):56-87. doi: 10.1016/S1474-4422(18)30415-0. Epub 2018 Nov 26. PMID 30497965
- [Derived] Mm P, Lg A, E G, C P, Mem B, Rjr F, Rm M, Af C, Jmd G, A A, B S, N M, K J, H C, Ga L. Time Course of Motor Improvement by Epidural Stimulation After Spinal Cord Injury: An Interim Analysis of a Phase II Trial. J Cent Nerv Syst Dis. 2025 Sep 22;17:11795735251379220. doi: 10.1177/11795735251379220. eCollection 2025. PMID 40994969